CLINICAL TRIAL: NCT06924190
Title: Clinical Equivalency Study of Two Formulations of Budesonide Inhalation Aerosol
Brief Title: Pharmacokinetics and Bioequivalence Study of Budesonide Inhalation Aerosol in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lunan Better Pharmaceutical Co., LTD. (Industry)
Collaborators: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BT-BDND-IA-BE01
Record Dates: First submitted 2025-03-29; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Bioequivalence Study in Healthy Subjects
Keywords: Budesonide Inhalation Aerosol
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference Group [Budiair® 200ug/puff ( budesonide inhalation aerosol )] (Active Comparator): After being trained and qualified, the subjects strictly administered one puff （Budiair®，200ug/puff ）of the investigational drug under the supervision of the investigator in accordance with the SOP for drug administration. After taking the medication, the subjects thoroughly rinsed their mouths multiple times with 150 mL of water and then spat out the mouthwash.
  Interventions: Drug: Budiair® 200ug/puff inhalation aerosol
- Test Group [200ug/puff (budesonide inhalation aerosol)] (Experimental): After being trained and qualified, the subjects strictly administered one puff （budesonide inhalation aerosol，200ug/puff ）of the investigational drug under the supervision of the investigator in accordance with the SOP for drug administration. After taking the medication, the subjects thoroughly rinsed their mouths multiple times with 150 mL of water and then spat out the mouthwash.
  Interventions: Drug: budesonide 200ug/puff inhalation aerosol

INTERVENTIONS:
Drug: Budiair® 200ug/puff inhalation aerosol — The subjects randomly received one puff Budiair®(budesonide inhalation aerosol 200ug/puff )
  Other Names: Budiair®
  Arms: Reference Group [Budiair® 200ug/puff ( budesonide inhalation aerosol )]
Drug: budesonide 200ug/puff inhalation aerosol — The subjects randomly received one puff budesonide inhalation aerosol(200ug/puff )
  Arms: Test Group [200ug/puff (budesonide inhalation aerosol)]

SUMMARY:
The test formulation of Budesonide Inhalation Aerosol is bioequivalent to the reference formulation in healthy Chinese subjects under fasting conditions.

DETAILED DESCRIPTION:
In a four-period single-dose oropharyngeal inhalation study of the investigational drug, with a washout period of 3 days. After dosing, subjects should thoroughly rinse their mouth with 150 ml of water and spit out the rinse water.

Blood plasma concentrations of budesonide are collected within the specified sampling time for pharmacokinetic parameter analysis. In each period, blood samples are collected at pre-dose 0 h and at 0.03, 0.07, 0.10, 0.13, 0.17, 0.20, 0.25, 0.33, 0.42, 0.50, 0.75, 1, 2, 4, 6, 8, 10, 12, and 16 h post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. **Age**: Chinese male or female subjects aged 18 to 65 years (inclusive of the boundary values).
2. **Weight**: Males must weigh ≥50.0 kg, and females must weigh ≥45.0 kg. The Body Mass Index (BMI) calculated as \[ \text{BMI} = \frac{\text{weight (kg)}}{\text{height}^2 (\text{m}^2)} \] must be between 19.0 and 26.0 kg/m² (inclusive of the boundary values).
3. **Informed Consent**: Subjects must fully understand the purpose, nature, methods, and potential adverse reactions of the trial and voluntarily sign a written informed consent form.
4. **Communication and Compliance**: Subjects must be able to communicate effectively with the investigator, correctly use the inhaler device after training, and understand and comply with all the requirements of the study.

Exclusion Criteria:

1. **Examination**: Subjects with clinically significant abnormalities in physical examination, vital signs, ECG, chest X-ray, complete blood count, urinalysis, or biochemical blood tests; subjects with serum potassium levels below the lower limit of normal.
2. **Examination**: Subjects with positive test results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), human immunodeficiency virus antigen and antibody (HIV), or syphilis antibody.
3. **Examination**: Subjects with a measured FEV1/predicted FEV1 ≤ 80% or FVC ≤ 80% of the predicted value in pulmonary function tests; or subjects whose pulmonary function test results are judged by the investigator to indicate small airway disease.
4. **Inquiry**: Subjects with a history or current diagnosis of chronic or severe diseases of the liver, kidneys, endocrine system, urinary system, digestive system, blood, or lymphatic system.
5. **Inquiry**: Subjects with a history or current diagnosis of chronic or severe respiratory diseases.
6. **Inquiry**: Subjects with a history or current diagnosis of chronic or severe cardiovascular diseases (especially ischemic heart disease, hypertension, aneurysm, paroxysmal tachycardia, etc.).
7. **Inquiry**: Subjects with a history or current diagnosis of chronic or severe nervous system diseases; or subjects with a history of frequent headaches or dizziness, or those who have experienced headaches or dizziness within one week before screening.
8. **Inquiry**: Subjects with a history of allergy to budesonide, its excipients, or other corticosteroid components; or subjects with a known history of allergies to two or more food or environmental substances, or a history of atopic allergic diseases (urticaria, rash, eczematous dermatitis, etc.).
9. **Inquiry**: Subjects with a history or current diagnosis of glaucoma, cataracts, or blurred vision.
10. **Examination**: Subjects with current oral ulcers, pharyngitis, or enlarged tonsils.
11. **Inquiry**: Subjects who consumed excessive amounts of tea, coffee, or caffeine-containing beverages (8 cups or more per day, 1 cup = 250 mL) within three months before screening, or those who do not agree to abstain from these beverages during the trial.
12. **Inquiry**: Subjects who consumed food that may affect drug metabolism (including grapefruit or grapefruit products, dragon fruit, mango, pomelo, etc.) within 48 hours before screening, or those who do not agree to abstain from such food during the trial.
13. **Inquiry**: Subjects with special dietary requirements that prevent adherence to a uniform diet, or those with difficulty swallowing.
14. **Inquiry + Examination**: Subjects who cannot tolerate venipuncture or have a history of fainting due to blood or needles, or those with difficulty in blood collection.
15. **Inquiry**: Subjects who have undergone surgery that the investigator judges may affect drug absorption, distribution, metabolism, or excretion; or those who plan to undergo surgery within four weeks before screening or during the trial.
16. **Inquiry**: Subjects who used any medication (prescription drugs, over-the-counter drugs, health supplements, vaccines, herbal medicines, etc.) within 30 days before screening.
17. **Examination**: Subjects with a positive alcohol breath test result (breath alcohol content > 0.0 mg/100 mL).
18. **Inquiry**: Subjects with a history of alcohol abuse within the past year (consuming ≥14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine) or those who cannot abstain from alcohol during the trial.
19. **Inquiry**: Subjects who smoked ≥5 cigarettes per day within three months before screening or those who cannot quit smoking during the trial.
20. **Examination**: Subjects with a positive urine nicotine test result.
21. **Inquiry + Internet Screening**: Subjects who participated in any drug clinical trial within three months before screening and received medication, or those who plan to participate in other clinical trials during this study.
22. **Inquiry**: Subjects who donated blood or had significant bleeding (more than 400 mL) within three months before screening; or those who plan to donate blood or blood components during the study or within three months after the study ends.
23. **Examination**: Subjects with a positive urine drug abuse screening result.
24. **Inquiry**: Subjects with a history of drug abuse within the past five years.
25. **Inquiry + Examination**: Pregnant or breastfeeding women, or women of childbearing age who had unprotected sexual intercourse with their partners within 14 days before screening.
26. **Inquiry**: Female subjects who used long-acting estrogen or progesterone injections or implants within six months before screening.
27. **Inquiry**: Male subjects (or their partners) or female subjects who plan to conceive or donate sperm or eggs during the entire trial period and within three months after the study ends, and are unwilling to take appropriate contraceptive measures.
28. Subjects with poor compliance.
29. Subjects who may not be able to complete the study for other reasons, or those whom the investigator deems unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Chinese male or female subjects
Enrollment: 32 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 12 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 12 days
  plasma concentration-time curve from zero to the time of the last measurable time point t
Area under the plasma concentration versus time curve (AUC)0-∞ | 12 days
  area under the plasma concentration-time curve from zero to infinity

OTHER OUTCOMES:
maximum plasma concentration (tmax) | 12 days
  time to reach the maximum plasma concentration after drug administration (tmax)
Incidence of Treatment-Emergent Adverse Events | During 12 days
  Collection of adverse events
Incidence of abnormal blood pressure | During 12 days
  Monitor the blood pressure
Incidence of abnormal temperature | During 12 days
  Monitor the temperature
Incidence of abnormal pulse | During 12 days
  Monitor the pulse

CONTACTS AND LOCATIONS:
Overall Officials: Kai Huang, Dr, Principal Investigator — Wuxi People's Hospital
Locations (2):
- China (2):
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Lunan Better Pharmaceutical Co., Ltd., Linyi, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang K, Yin S, Huang W, Ding L, Qin W, Qian Z, Ding Y, Que L, Shi Y, Gao J, Zhao Y. A Single Dose, Randomized, Open-Label, Cross-Over Bioequivalence Study of Budesonide Pressurized Metered-Dose Inhaler in Healthy Chinese Subjects. Pharmacol Res Perspect. 2025 Dec;13(6):e70197. doi: 10.1002/prp2.70197. PMID 41318994